CLINICAL TRIAL: NCT05561803
Title: The Use of Photobiomodulation in the Management of Radiodermatitis in Patients in Palliative Care. A Prospective Study.
Status: Withdrawn | Type: Observational
Why Stopped: Research team withdrawn the study before starting the recruitment because the university suspended the service for administrative restructuring
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Rebeca Boltes Cecatto, Professor Rebeca Boltes Cecatto, University of Nove de Julho
Other Study IDs: Radiodermatitistalita30
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Radiodermatitis; Acute; Radiotherapy Side Effect; Cancer Patients; Palliative Care
Keywords: Radiodermatitits; Radiotherapy; Photobiomodulation; Cancer; Palliative Care
MeSH Terms: conditions — Radiodermatitis; Radiation Injuries; Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radiodermatitis Case Group: 40 patients on palliative care with grade 2 or grade 3 radiodermatitis after radiotherapy for the treatment of cancer submitted to a PBM therapy protocol
  Interventions: Radiation: Photobiomodulation Therapy

INTERVENTIONS:
Radiation: Photobiomodulation Therapy — Focal low-level laser therapy, Red Laser (wavelength 633 nm to 685 nm), or Infrared Laser Laser (wavelength 780 nm to 830 nm), with a low-intensity laser equipment of 100 mW and a cross-sectional area of the device beam of 0.0434 cm². The parameters are 1 to 3 J per point, with equidistant points of 1.5 to 2 cm, covering the entire length of the open lesion. Therapy is carried out every 48 hours until the total wound healing, regardless of the number of sessions required.
  Other Names: PBM Therapy

SUMMARY:
It is estimated that there will be 670,000 new cases of cancer worldwide in 2020-2022 and it is known that the most commonly instituted treatments in cancer are chemotherapy, radiotherapy and surgery. However, these treatments have undesirable side effects, such as Radiodermatitis after Radiotherapy (RD). In fact, the prevalence of possible side effects after radiotherapy is estimated to be 80 to 90%. Radiotherapy complications are associated with a negative impact on patients' quality of life and few supportive measures are available for such complications. Thus, the management of these side effects has been studied in the literature until the present day. On the other hand, Photobiomodulation (PBM) has an important role in wound repair and tissue regeneration, as it influences the different phases of lesion resolution, including the inflammatory phase, the proliferative phase and the remodeling phase. Thus, the aim of this study is to report a case series of Cancer Patients diagnosed with radiotherapy-induced acute radiodermatitis on Palliative Care, treated with PBM. This is a case series report and the study data will be extracted from the medical records of forty cancer patients with grade 2 or 3 RD followed up from September 2023 at the Laser Therapy Outpatient Clinic in a Universitary Hospital. The outcomes are the size of the lesion, the presence of pain assessed by the Visual Analogue Scale (VAS), the Portuguese Version of WHOQOL BREF Scale and the RTOG Scale (Radiation Therapy Oncology Group Scale) to assess the degree of Radiodermatitis before and after PBM therapy. The data will be subjected to a statistical analysis and will be discussed. Data with positive or negative results will be reported.

DETAILED DESCRIPTION:
It is estimated that there will be 670,000 new cases of cancer worldwide in 2020-2022 and it is known that the most commonly instituted treatments in cancer are chemotherapy, radiotherapy and surgery. However, these treatments have undesirable side effects, such as Radiodermatitis after Radiotherapy (RD). In fact, the prevalence of possible side effects after radiotherapy is estimated to be 80 to 90%. Radiotherapy complications are associated with a negative impact on patients' quality of life and few supportive measures are available for such complications. Thus, the management of these side effects has been studied in the literature until the present day. On the other hand, Photobiomodulation (PBM) has an important role in wound repair and tissue regeneration, as it influences the different phases of lesion resolution, including the inflammatory phase, the proliferative phase and the remodeling phase. Thus, the aim of this study is to report a case series of forty cancer patients on palliative care diagnosed with radiotherapy-induced acute radiodermatitis Grade 2or 3, treated with PBM. This is a case series report and the study data will be extracted from the medical records of patients with grade 2 or 3 RD followed up from September 2023 at the Laser Therapy Outpatient Clinic in a Universitary Hospital. The outcomes are the size of the lesion, the presence of pain assessed by the Visual Analogue Scale (VAS), the Portuguese Version of WHOQOL BREF Scale and the RTOG Scale (Radiation Therapy Oncology Group Scale) to assess the degree of Radiodermatitis before and after PBM therapy. The assessment will be done pre-treatment, weekly during PBM therapy and post-treatment. The PBM therapy are focal low-level laser therapy, 1 to 3 Joules per point, depending on the degree of pain, wavelength 633 to 685 nm, transcutaneously on the surface of the tissue injured by radiotherapy, three times a week during radiotherapy treatment and two more applications after the end of radiotherapy The data will be subjected to a statistical analysis and will be discussed. Data with positive or negative results will be reported.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years;
2. Patients with any oncological etiology;
3. With the presence of established radiodermatitis RTOG II or III;
4. Patients who are undergoing palliative oncological care and RD standard treatment;
5. Patients who do not present clinical signs of another pathology that justifies the presence of the skin lesion;
6. Patients do not have local skin infection

Exclusion Criteria:

* Critical clinical states;
* Patients with skin lesions of another cause even when undergoing RT;
* Patients referred to the laser clinic for the prevention of radiodermatitis without the active RD lesion.
* Patients who have used another photobiomodulation therapy protocol foresaw injury not related to the study.
* All contraindications already defined in the routine referral to the outpatient clinic (patients who have an active tumor at the site to be irradiated; individuals with a history of photosensitivity to photonic or light therapy; patients who have undiagnosed lesions in the treatment region; patients using topical photosensitizing medications or creams; cognitive, psychiatric or neurological changes that prevent the free understanding of the PBM therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatient cancer patients on palliative care undergoing radiotherapy and who show signs of radiodermatitis RTOG II OR III.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-04-08 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Toxicity criteria of the Radiation Therapy Oncology Group Scale (RTOG Scale) | Change from Baseline at 14 days after end of radiotherapy treatment]
  RTOG scale assess the degree and intensity of RD. It identifies degree 0 (no reaction), 1 (faint erythema, dry desquamation, epilation, diminished sweating), 2 (moderate, brisk erythema, exudative dermatitis in plaques and moderate edema), 3 (exudative dermatitis, besides cutaneous folds and intense edema) and 4 (ulceration, hemorrhage, necrosis).
Lesion Size | Change from Baseline at 14 days after end of radiotherapy treatment]
  Evaluation of lesion measurement in centimeters
Portuguese version of The World Health Organization Quality of Life Scale (WHOQOL-BREF) | Change from Baseline at 14 days after end of radiotherapy treatment]
  The WHOWOL BREF scale assess multidimensional aspects of geral quality of life of patients. The multidimensional scale is composed by 26 items, classified from 1 to 5 according to the intensity of the symptom presented. The global score is calculated by adding up all the items as well as the score for each domain is evaluated adding it individually for each item, which can range from 0 to 130,

SECONDARY OUTCOMES:
Visual Analog Scale of Pain | Change from Baseline at 14 days after end of radiotherapy treatment]
  VAS Scale assess the pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

CONTACTS AND LOCATIONS:
Overall Officials: Rebeca B Cecatto, Ph.D., Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho / Post-Graduate program Biophotonics Applied to Health Sciences, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No